CLINICAL TRIAL: NCT00304941
Title: Breast Cancer and Insulin Resistance: Implications for Preventive Counseling in Familial and Sporadic Cases
Brief Title: Insulin Resistance and Breast Cancer
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060119; 06-CH-0119
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-17

CONDITIONS: Breast Cancer; Insulin Resistance
Keywords: Breast Cancer; Family History; Pre/Post Menopausal; Prevention; Risk-Factor; Body-Mass-Index; BRCA1; Insulin; Genetic Counseling; Penetrance; Risk Assessment; Healthy Volunteer; HV
MeSH Terms: conditions — Breast Neoplasms; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will characterize risk factors associated with breast cancer development in some patients. In particular, it will examine the role of insulin in breast cancer in patients with and without a family history of the disease.

Women 30 to 70 years old who have been diagnosed with breast cancer and matched control healthy subjects with and without a family history of breast cancer may be eligible for this study.

Participants undergo the following procedures:

* Cancer-genetic counseling session, including family history, risk assessment, genetic testing for BRCA1 and BRCA2 (if criteria is met), interpretation of results and management options
* Medical history, including questions about symptoms or diseases, reproductive history, use of oral contraceptives, body weight, exercise, lifestyle, and demographic issues
* Drawing of family tree
* Examination of medical records
* Blood drawing for genetic and other tests
* CT scan of the abdomen (approximate time < 1 minute)
* Filling out questionnaires

DETAILED DESCRIPTION:
The etiology of breast cancer is still poorly understood with known risk factors explaining only a small proportion of cases. Risk factors that modulate the development of breast cancer include: age, geographic location, socioeconomic status, reproductive events, exogenous hormones, lifestyle, familial history of breast cancer, mammographic density, history of benign breast disease, ionizing radiation, and bone density.

Several lines of evidence have demonstrated that insulin and the insulin receptor play a key role in the formation and progression of breast cancer. Insulin has direct and indirect effects on breast cancer; direct effects as a growth promoting factor and indirect effects through actions on other hormones involved in breast cancer. In addition, certain conditions associated with insulin resistance, such as obesity and abdominal fat, are known risk factors for breast cancer.

Family history of breast cancer is also a well established major risk factor. To date, both genetic and non-genetic factors have been suggested to influence breast cancer risk in women with a positive family history of breast cancer including those with recognized mutations in the BRCA1 and BRCA2 genes. Women with a family history of breast cancer inherit a susceptibility to the condition; the development of the disease requires a series of promoting steps including lifestyle, diet, and environmental factors. Several hormones involved in breast cancer such as IGF-1, testosterone, and SHBG are affected by a positive family history of breast cancer. Also, women with a high Waist-to-Hip ratio (WHR) and a positive family history of breast cancer are at higher risk of developing breast cancer than those women with a high WHR without a positive family history. The role of insulin and insulin-related factors in women with a family history of breast cancer has not been examined.

There is growing recognition that insulin may be a potential mediator of breast cancer. The above evidence suggests that actions of insulin may be involved in the promoting steps that predispose some women to breast cancer. These findings provide the biological basis for insulin related factors to serve as potential targets for breast cancer prevention and risk assessment.

The main goal of this proposal is to unravel the contributions of insulin and insulin-related actions (e.g. insulin resistance, abdominal fat) on breast cancer risk. The purpose of the present study is to characterize the role of insulin in newly diagnosed premenopausal and postmenopausal women with and without a family history of breast cancer. The objective is to assess the relative strength of each risk factor associated with insulin actions and their individual impact on breast cancer. This study will provide data that may serve as the basis for future studies on preventive strategies targeted at lowering insulin levels and increasing insulin sensitivity (e.g. decrease glucose, decrease abdominal fat, decrease omega-6 fatty acids/increase omega-3 fatty acids, increase fiber intake, increase exercise) in a subset of patients.

This protocol will recruit only female patients, and will concentrate only on breast cancer risk. Subjects will be asked to complete several questionnaires in the course of genetic counseling to provide information on medical and reproductive history, demographics, risk factors, physical activity as well as other information needed to establish an appropriate sample for the study. Genetic testing will be offered as part of the initial evaluation and to check for BRCA1/2 mutation status.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Females (ages 30-70 years old) who have been diagnosed with breast cancer and age matched controls with and without a family history of breast cancer.

The actual selection of patients most appropriate for research and clinical training needs will be made by protocol investigators.

Referrals will be accepted from the patient recruitment office of the NIH, genetic counselors, geneticists, oncologists, and other health care providers in the area or anybody who reads the information about the study on the NIH world wide web site.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-03-14; Study Completion 2010-09-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dumitrescu RG, Cotarla I. Understanding breast cancer risk -- where do we stand in 2005? J Cell Mol Med. 2005 Jan-Mar;9(1):208-21. doi: 10.1111/j.1582-4934.2005.tb00350.x. PMID 15784178
- [Background] Wolf I, Sadetzki S, Catane R, Karasik A, Kaufman B. Diabetes mellitus and breast cancer. Lancet Oncol. 2005 Feb;6(2):103-11. doi: 10.1016/S1470-2045(05)01736-5. PMID 15683819
- [Background] Milazzo G, Giorgino F, Damante G, Sung C, Stampfer MR, Vigneri R, Goldfine ID, Belfiore A. Insulin receptor expression and function in human breast cancer cell lines. Cancer Res. 1992 Jul 15;52(14):3924-30. PMID 1617668